CLINICAL TRIAL: NCT03058640
Title: The Effects of Participation in Karate on Health Outcomes in Adolescents With Down Syndrome
Brief Title: Effects of Karate in Adolescents With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Down Syndrome Association of Toledo (Unknown)
Responsible Party: Principal Investigator, Dale A Ulrich, Professor of Physical Education and Movement Science, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00116460
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Karate Intervention (Experimental): Participants will be enrolled into PKSA karate classes which includes at least two, standardized 1-hour classes per week for 12 weeks. Participants must attend at LEAST 20/24 classes. Attendance sheets will be signed by parents at each site. Practice at home will also be encouraged. Log sheets will be provided to participants to log their practice
  Interventions: Other: PKSA karate class
- Standard Care (No Intervention): Participants will have no initial intervention. Investigators will request that participants do not enroll in a structured martial arts class during the one-year period. Participants will, however, be given the option of receiving the structured karate program at 6 months, once measurements are completed

INTERVENTIONS:
Other: PKSA karate class — Participants will attend at least 20/24 PKSA karate classes over a 12 week period, completing standard karate training lessons. Participants will also be encouraged to practice on their own at home.
  • Participants must attend at LEAST 20/24 classes
  Arms: Karate Intervention

SUMMARY:
This randomized control study will investigate the health outcomes of adolescents with Down Syndrome who participate in a karate class as measured by ALPHA fitness testing and various PROMIS parent proxy questionnaires to assess participants mobility, physical activity, and overall affect.

DETAILED DESCRIPTION:
Adolescents with Down syndrome suffer from a set of health problems including heart disease, sleep disturbances, and obesity. Their decreased cardiovascular fitness and exercise capacity limits their ability to perform activities of daily living. Exercise interventions in this population of children have been shown to improve muscle strength, balance, and cardiovascular fitness. Prior research has helped better define physical activity barriers in this population which include: requiring parental supervision, lack of accessible programs, seasonal activities and reduced physical skills of the child. Karate is an indoor activity that can be performed at different skill levels without parental involvement. The investigators hypothesize that adolescents with Down syndrome who participate in karate will show improved health outcomes compared to those who did not participate. Furthermore, the investigators hypothesize that the majority of participants will continue the activity outside of the research window. This randomized controlled trial will enroll 30 adolescents with Down syndrome. Participants will be randomly assigned to a 3 month karate program or the control group with no intervention. Measurements are taken at baseline, 3 months, and 6 months using validated ALPHA fitness testing and in addition parents will complete PROMIS questionnaires to assess overall participant's activity level, mobility, and generalized affect. An independent statistician will analyze the groups. This research will help physicians provide adolescents with Down syndrome appropriate recommendations for an individualized physical activity regimen that does not have similar limitations to other exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* males & females with a diagnosis of down syndrome
* Ability to participate in 2 hours of exercise per week
* No involvement in formal martial arts classes over the past 3 months

Exclusion Criteria:

* Behavior problems that would prevent them from participating in organized classes
* Health problems that preclude them from participating in moderate physical activity programs (e.g. uncontrolled seizures)
* No Co-existing diagnosis (e.g. ASD)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Balance | Measure difference between baseline and three months
  Will measure the length of time that participant can stand on one foot (up to 30 seconds)
20m shuttle run | Measure difference between baseline and three months
  Participants are to run between 2 lines, 20 m apart in time with an audio signal. The speed of the signal is increased by 0.5 km/h/min. The test finishes when the participant fails to reach the end lines concurrent with audio signals on 2 consecutive occasions (or when participant stops because of fatigue)
standing long jump | Measure difference between baseline and three months
  measure length of distance jumped from static position as part of Alpha Fitness Test
handgrip strength | Measure difference between baseline and three months
  Squeeze hand dynamometer as hard as possible for seconds. This will be repeated with both hands twice
tricep skin fold test | Measure difference between baseline and three months
  Width of skin fold test as measured with calipers as part of Alpha Fitness Test
waist circumference | Measure difference between baseline and three months
  Simple measure of waist circumference as part of Alpha Fitness Test
BMI | Measure difference between baseline and three months
  Calculation of body mass index by taking participants weight in kg divided by height in meters squared
PROMIS Parent Proxy Mobility SF v.2.0 - | Measure difference between baseline and three months
  Parent completed questionnaire including eight questions that gauges parent confidence that their child could perform various mobility related tasks with "no trouble", "a little trouble", "some trouble", "a lot of trouble", or "not able to do"
PROMIS Parent Proxy Physical Activity SF v1.0 | Measure difference between baseline and three months
  Parent completed questionnaire including eight questions that gauges parent's perception of how often their child was able to perform physical activity/exercise over the course of the seven days prior to completing the questionnaire
PROMIS Parent Proxy Positive Affect SF v1.0 | Measure difference between baseline and three months
  Parent completed questionnaire including eight questions that gauges parent's perception of how often their child felt happy, great, cheerful, joyful, in a good mood, refreshed, calm, peaceful

SECONDARY OUTCOMES:
Balance | Measure difference between baseline and 6 months
  Will measure the length of time that participant can stand on one foot (up to 30 seconds)
20m shuttle run | Measure difference between baseline and 6 months
  Participants are to run between 2 lines, 20 m apart in time with an audio signal. The speed of the signal is increased by 0.5 km/h/min. The test finishes when the participant fails to reach the end lines concurrent with audio signals on 2 consecutive occasions (or when participant stops because of fatigue)
standing long jump | Measure difference between baseline and 6 months
  measure length of distance jumped from static position as part of Alpha Fitness Test
handgrip strength | Measure difference between baseline and 6 months
  Squeeze hand dynamometer as hard as possible for seconds. This will be repeated with both hands twice
tricep skin fold test | Measure difference between baseline and 6 months
  Width of skin fold test as measured with calipers as part of Alpha Fitness Test
waist circumference | Measure difference between baseline and 6 months
  Simple measure of waist circumference as part of Alpha Fitness Test
BMI | Measure difference between baseline and 6 months
  Calculation of body mass index by taking participants weight in kg divided by height in meters squared
PROMIS Parent Proxy Mobility SF v.2.0 - | Measure difference between baseline and 6 months
  Parent completed questionnaire including eight questions that gauges parent confidence that their child could perform various mobility related tasks with "no trouble", "a little trouble", "some trouble", "a lot of trouble", or "not able to do"
PROMIS Parent Proxy Physical Activity SF v1.0 | Measure difference between baseline and 6 months
  Parent completed questionnaire including eight questions that gauges parent's perception of how often their child was able to perform physical activity/exercise over the course of the seven days prior to completing the questionnaire
PROMIS Parent Proxy Positive Affect SF v1.0 | Measure difference between baseline and 6 months
  Parent completed questionnaire including eight questions that gauges parent's perception of how often their child felt happy, great, cheerful, joyful, in a good mood, refreshed, calm, peaceful

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hornyak, MD, Principal Investigator — University of Michigan PM&R; Dale Ulrich, PhD, Principal Investigator — University of Michigan School of Kinesiology
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr M, Shields N. Identifying the barriers and facilitators to participation in physical activity for children with Down syndrome. J Intellect Disabil Res. 2011 Nov;55(11):1020-33. doi: 10.1111/j.1365-2788.2011.01425.x. Epub 2011 May 10. PMID 21554468
- [Background] Chen CC, Ringenbach SD, Crews D, Kulinna PH, Amazeen EL. The association between a single bout of moderate physical activity and executive function in young adults with Down syndrome: a preliminary study. J Intellect Disabil Res. 2015 Jul;59(7):589-98. doi: 10.1111/jir.12163. Epub 2014 Aug 29. PMID 25171600
- [Background] Cowley PM, Ploutz-Snyder LL, Baynard T, Heffernan K, Jae SY, Hsu S, Lee M, Pitetti KH, Reiman MP, Fernhall B. Physical fitness predicts functional tasks in individuals with Down syndrome. Med Sci Sports Exerc. 2010 Feb;42(2):388-93. doi: 10.1249/MSS.0b013e3181b07e7a. PMID 19927019
- [Background] Shields N, Dodd KJ, Abblitt C. Do children with Down syndrome perform sufficient physical activity to maintain good health? A pilot study. Adapt Phys Activ Q. 2009 Oct;26(4):307-20. doi: 10.1123/apaq.26.4.307. PMID 19893069
- [Background] Andriolo RB, El Dib RP, Ramos L, Atallah AN, da Silva EM. Aerobic exercise training programmes for improving physical and psychosocial health in adults with Down syndrome. Cochrane Database Syst Rev. 2010 May 12;2010(5):CD005176. doi: 10.1002/14651858.CD005176.pub4. PMID 20464738
- [Background] Elmahgoub SS, Van de Velde A, Peersman W, Cambier D, Calders P. Reproducibility, validity and predictors of six-minute walk test in overweight and obese adolescents with intellectual disability. Disabil Rehabil. 2012;34(10):846-51. doi: 10.3109/09638288.2011.623757. Epub 2011 Dec 10. PMID 22149772
- [Background] Izquierdo-Gomez R, Martinez-Gomez D, Acha A, Veiga OL, Villagra A, Diaz-Cueto M; UP&DOWN study group. Objective assessment of sedentary time and physical activity throughout the week in adolescents with Down syndrome. The UP&DOWN study. Res Dev Disabil. 2014 Feb;35(2):482-9. doi: 10.1016/j.ridd.2013.11.026. Epub 2013 Dec 25. PMID 24374601
- [Background] Lotan M. Quality physical intervention activity for persons with Down syndrome. ScientificWorldJournal. 2007 Jan 10;7:7-19. doi: 10.1100/tsw.2007.20. PMID 17221138
- [Background] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus JA. Physical activity and cardiorespiratory fitness in adolescents with Down syndrome. Nutr Hosp. 2013 Jul-Aug;28(4):1151-5. doi: 10.3305/nh.2013.28.4.6509. PMID 23889635
- [Background] Mendonca GV, Pereira FD, Fernhall B. Reduced exercise capacity in persons with Down syndrome: cause, effect, and management. Ther Clin Risk Manag. 2010 Dec 8;6:601-10. doi: 10.2147/TCRM.S10235. PMID 21206759
- [Background] Pikora TJ, Bourke J, Bathgate K, Foley KR, Lennox N, Leonard H. Health conditions and their impact among adolescents and young adults with Down syndrome. PLoS One. 2014 May 12;9(5):e96868. doi: 10.1371/journal.pone.0096868. eCollection 2014. PMID 24818963
- [Background] Tejero-Gonzalez CM, Martinez-Gomez D, Bayon-Serna J, Izquierdo-Gomez R, Castro-Pinero J, Veiga OL. Reliability of the ALPHA health-related fitness test battery in adolescents with Down syndrome. J Strength Cond Res. 2013 Nov;27(11):3221-4. doi: 10.1519/JSC.0b013e31828bed4e. PMID 23442277
- [Background] Vis JC, de Bruin-Bon RH, Bouma BJ, Backx AP, Huisman SA, Imschoot L, Mulder BJ. 'The sedentary heart': physical inactivity is associated with cardiac atrophy in adults with an intellectual disability. Int J Cardiol. 2012 Jul 26;158(3):387-93. doi: 10.1016/j.ijcard.2011.01.064. Epub 2011 Feb 26. PMID 21353712
- [Background] Vis JC, Thoonsen H, Duffels MG, de Bruin-Bon RA, Huisman SA, van Dijk AP, Hoendermis ES, Berger RM, Bouma BJ, Mulder BJ. Six-minute walk test in patients with Down syndrome: validity and reproducibility. Arch Phys Med Rehabil. 2009 Aug;90(8):1423-7. doi: 10.1016/j.apmr.2009.02.015. PMID 19651279
- [Background] Casey AF, Wang X, Osterling K. Test-retest reliability of the 6-minute walk test in individuals with Down syndrome. Arch Phys Med Rehabil. 2012 Nov;93(11):2068-74. doi: 10.1016/j.apmr.2012.04.022. Epub 2012 May 7. PMID 22575394